CLINICAL TRIAL: NCT04981821
Title: A Pilot Randomized Trial of a Mobile Health Exercise Intervention for Older Patients With Myeloid Neoplasms
Brief Title: A Randomized Trial of a Mobile Health Exercise Intervention for Older Adults With Myeloid Neoplasms
Acronym: GO-EXCAP2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kah Poh Loh, Assistant Professor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCS21043; R00CA237744 (NIH)
Record Dates: First submitted 2021-07-27; First posted 2021-07-29 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Myeloid Neoplasm
Keywords: mobile health exercise intervention; Myeloid Neoplasm; GO-EXCAP
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GO-EXCAP (Experimental): GO-EXCAP Mobile App involves the use of a mobile app delivery platform to deliver an exercise program [Exercise for Cancer Patients (EXCAP©®)]. EXCAP©®) is a progressive walking and resistance exercise program
  Interventions: Behavioral: GO-EXCAP Mobile App
- Behavioral Placebo Control (Active Comparator): Participants will meet with an oncology nurse (for approximately 60 min) to review the NCI booklet Chemotherapy and You: Support for People With Cancer, which includes facts about chemotherapy and its side effects. They will be provided with NCI online resources to review at home.
  Interventions: Behavioral: Behavioral Placebo Control

INTERVENTIONS:
Behavioral: GO-EXCAP Mobile App — A mobile app delivery platform to deliver an exercise program [Exercise for Cancer Patients (EXCAP©®)]. EXCAP©®) is a progressive walking and resistance exercise program
  Arms: GO-EXCAP
Behavioral: Behavioral Placebo Control — Participants will meet with an oncology nurse (for approximately 60 min) to review the NCI booklet Chemotherapy and You: Support for People With Cancer, which includes facts about chemotherapy and its side effects. They will be provided with NCI online resources to review at home.
  Arms: Behavioral Placebo Control

SUMMARY:
This is a phase 2 randomized controlled trial (RCT) to assess the preliminary efficacy of the a mobile health exercise intervention (GO-EXCAP) versus a chemotherapy education control in 100 older patients with MN receiving outpatient chemotherapy on physical function and patient-reported outcomes (fatigue, mood, and quality of life). We will also explore the effect of the intervention on TNFα and related cytokine gene promoter methylation and their gene and protein expression.

DETAILED DESCRIPTION:
Up to 98% of older patients with myeloid neoplasms experience physical function decline, fatigue, and mood disturbances. Mobile health exercise interventions are promising strategy to prevent physical function decline and improve fatigue and mood disturbances, but older patients with myeloid neoplasms receiving outpatient chemotherapy are understudied. The proposed study will investigate whether a novel mobile health exercise intervention that is adapted to this population can prevent physical function decline, improve fatigue and mood disturbances, and prevent worsening quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years (conventional definition of older age in clinical trials of MN)
* Have a diagnosis of MN
* Planned for or receiving outpatient cancer-directed treatments (participants receiving consolidative or maintenance outpatient therapies after induction chemotherapy are allowed to enroll)
* English speaking
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* No medical contraindications for exercise per oncologist
* Able to walk 4 meters as part of Short Physical Performance Battery measured walk (with or without assistive device)
* Able to provide informed consent

Exclusion Criteria:

* Physical, psychological, or social impairments that would interfere with subject's ability to participate in the study or participate in the intervention, as determined by the PI or the treating team

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference between experimental and active comparator arms- Physical Function | 12 Weeks
  Changes in physical function measured using the Short Physical Performance Battery (SPPB) which an objective physical assessment evaluating lower extremity physical function (score ranges from 0-12; higher score indicates better physical function). It is comprised of 3 components: a four-meter walk, repeated chair stands and a balance test (the score for each component ranges from 0-4).

SECONDARY OUTCOMES:
Difference between experimental and active comparator arms -Fatigue | 12 Weeks
  Changes in fatigue measures using the Brief Fatigue Inventory (BFI) which is a 9-item, patient-reported instrument. The score for each item ranges from 0-10, a higher score indicates higher self-reported levels of fatigue.
Difference between experimental and active comparator arms -Depression | 12 Weeks
  Changes in depression measured using the Center for Epidemiological Studies Depression Scale (CES-D) which is a 20-item depression scale. The score for each item ranges from 0-3, a higher score indicates higher self-reported depression levels.
Difference between experimental and active comparator arms -Quality of Life | 12 Weeks
  Changes in quality of life measured using the Functional Assessment of Cancer Therapy-Leukemia (FACT-Leu) scale. It consists of 44 items divided into 5 subscales: physical well-being (PWB), social well-being (SWB), emotional well-being (EWB), functional well-being (FWB) and leukemia-specific concerns. The score for each item ranges from 0-4. After reversing the scoring of negatively worded items, all the scores are summated. A higher score indicates better quality of life.

OTHER OUTCOMES:
Difference between experimental and active comparator arms -Inflammatory cytokines | 12 Weeks
  Inflammatory cytokines including TNFα, sTNFR1, sTNFR2, IL-1β, IL-2, IL-6, sIL-6R, IL-8, IL-10
Difference between experimental and active comparator arms- DNA methylation in the TNFα promoter region | 12 Weeks
  DNA methylation in the TNFα promoter region
Difference between experimental and active comparator arms- TNFα gene expression | 12 Weeks
  TNFα gene expression by PCR

CONTACTS AND LOCATIONS:
Overall Officials: Kah Poh Loh, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center/Wilmot Cancer Institute, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete and final study protocol will be made publicly available through the University of Rochester Cancer Center Community Oncology Research Program Research Base Protocol and Data Sharing Committee. The full protocol and data will be made publicly available no later than the publication date of the study findings from the final dataset. The protocol will include a detailed description of the study population, hypotheses tested, measurement and assessment information, data definitions and codes, and the analysis plan utilized. We will also make this protocol available to NIH and NCI at the time of submission of each progress report and at the end of the final funding year. We will be collecting identifying information. The final dataset will be stripped of identifiers prior to release for sharing.Published papers will be made available in portable document format.
Supporting Information: Study Protocol
Time Frame: The data will be available for 7 years after study completion.

REFERENCES:
- [Derived] Loh KP, Sanapala C, Jensen-Battaglia M, Rana A, Sohn MB, Watson E, Gilmore N, Klepin HD, Mendler JH, Liesveld J, Huselton E, LoCastro M, Susiarjo M, Netherby-Winslow C, Williams AM, Mustian K, Vertino P, Janelsins MC. Exercise and epigenetic ages in older adults with myeloid malignancies. Eur J Med Res. 2023 May 30;28(1):180. doi: 10.1186/s40001-023-01145-z. PMID 37254221